CLINICAL TRIAL: NCT03663348
Title: NYU Takotsubo (Broken Heart Syndrome) Registry
Brief Title: Registry of Patients With Takotsubo Syndrome
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 09-0746
Record Dates: First submitted 2018-05-16; First posted 2018-09-10 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Takotsubo Cardiomyopathy; Broken Heart Syndrome; Tako-tsubo Cardiomyopathy
MeSH Terms: conditions — Takotsubo Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Takotsubo syndrome is a condition which mimics acute myocardial infarction, and is diagnosed in 1.5% to 2.2% of patients referred to hospital with suspected acute coronary syndrome. It is also known as broken heart syndrome, takotsubo cardiomyopathy, stress cardiomyopathy and apical ballooning cardiomyopathy, among other names. The pathogenesis of this disorder is not well understood. Possible mechanisms include catecholamine excess, coronary artery spasm, microvascular dysfunction, among others. This is a multicenter, nation-wide, observational study of patients who were previously diagnosed with takotsubo syndrome. The investigators aim to use this registry to help plan and carry out further studies and to improve understanding of the pathophysiologic mechanisms of this syndrome. In addition participants will be followed for events, and to monitor quality of life and stress.

DETAILED DESCRIPTION:
Patients are eligible to participate if they are aged 18 years or older and carry a physician confirmed diagnosis of takotsubo syndrome. Patients with a history of takotsubo syndrome will be identified via physician referral, Epic search and patient self-referral. Patients may register directly through our registry website at www.nyulmc.org/brokenheartstudy or via direct contact with the study team via e-mail or telephone. Following completion of a research authorization form and collection of medical records, study team will confirm the diagnosis of takotsubo syndrome. Data will be collected including contact information, medical history, data on the takotsubo event(s) including physician records and all relevant imaging. Participants will also be asked quality of life questionnaires and will be followed every 4 months for events.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of takotsubo syndrome
* Age>18 years

Exclusion Criteria:

- Lack of capacity to provide informed consent

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with history of takotsubo syndrome
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-09-11 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events | up to 10 years
  Medical record review and patient report of repeat takotsubo event, MI, heart failure, unstable angina, chest pain ER visit, cardiovascular death, stroke

SECONDARY OUTCOMES:
Quality of life assessed using the Patient Reported Outcome Measurement Information System (PROMIS-10) questionnaire | every four months up to 10 years
  Measure of quality of life
Anxiety is assessed using the Hospital Anxiety and Depression Scale (HADS-A) | every four months up to 10 years
  Measure of anxiety
Depression assessed using the Patient Health Questionnaire (PHQ-9) | every four months up to 10 years
  Measure of depression
Perceived stress is measured using the Perceived Stress Scale (PSS-10) | every four months up to 10 years
  Measure of perceived stress

CONTACTS AND LOCATIONS:
Locations (1):
- NYU School of Medicine, New York, New York, United States